CLINICAL TRIAL: NCT03842137
Title: tDCS to Decrease Opioid Relapse
Brief Title: tDCS to Decrease Opioid Relapse (UG3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1810-001; UG3DA047793 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Opioid Dependence; Craving
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- tDCS (Active Comparator): Each participant will undergo 5 consecutive (i.e., business days) sessions of active tDCS delivered to the DLPFC. During each session, participants are engaging in tasks that activate the cognitive control network.
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): Each participant will undergo 5 consecutive (i.e., business days) sessions of sham tDCS delivered to the DLPFC. During each session, participants are engaging in tasks that activate the cognitive control network.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — Each participant will undergo 5 consecutive (i.e., business days) sessions of active tDCS delivered to the DLPFC. During each session, participants are engaging in tasks that activate the cognitive control network.
  Arms: tDCS
Device: sham tDCS — Each participant will undergo 5 consecutive (i.e., business days) sessions of sham tDCS delivered to the DLPFC. During each session, participants are engaging in tasks that activate the cognitive control network.
  Arms: sham tDCS

SUMMARY:
In the current proposal, the investigators will measure behavioral and brain responses following transcranial direct current stimulation (tDCS) to the dorsolateral prefrontal cortex (DLPFC) (anode on right DLPFC, cathode on the left DLPFC) delivered during cognitive control network (CCN) priming. Participants with opioid dependence, in the first month of prescribed buprenorphine or methadone, will be assessed twice using electroencephalographic (EEG), once prior to tDCS+CCN priming and again at the completion of 5 sessions of tDCS+CCN priming (one week later). EEG will provide validation of expected changes in these networks following tDCS stimulation of the DLPFC.

DETAILED DESCRIPTION:
Investigators propose to use EEG to examine oscillatory brain changes as well as self-reported craving before and after administration of five sessions of tDCS+Cognitive Control Network (CCN) priming stimulation vs. sham tDCS+CCN priming (randomized control trial) in 60 opioid dependent participants who recently initiated buprenorphine or methadone. Participants in the first month of prescribed buprenorphine or methadone will be assessed EEG, once prior to tDCS and again one week later after completion of 5 sessions of tDCS+CCN priming. EEG will be expected to provide 1) validation of expected network and oscillatory changes from tDCS-targeting and 2) an effect size for DLPFC vs sham stimulation. Go/no go criteria for the UG3 phase will be demonstration of enhanced frontal theta power during a WM task AND greater change (at least 10% difference between conditions, controlling for baseline craving) in subjective craving following the tDCS+CCN priming intervention compared to sham tDCS+CCN priming.

ELIGIBILITY:
Inclusion Criteria:

* current opioid dependence
* between 21-50 years of age
* recent initiation of buprenorphine or methadone (<30 days)

Exclusion Criteria:

* current criteria for a DSM-V diagnosis of bipolar disorder, schizophrenia, schizo-affective, schizophreniform, or paranoid disorder
* current suicidality
* evidence of neurocognitive dysfunction
* contraindications for tDCS (e.g seizure disorder)
* probation/parole requirements or an upcoming move that might interfere with protocol participation
* planning to terminate buprenorphine in less than 3 months
* scalp lesions near the tDCS electrode sites

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Abrantes, Ph.D., Principal Investigator — Butler Hospital; Michael D Stein, M.D., Principal Investigator — Boston University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment started June 4, 2019 and was completed on 2/21/23. Participants were recruited from both clinical settings and through community advertisements.
Pre-assignment Details: Once enrolled, participants were randomized at the beginning of their first tDCS session. If they did not attend that session, they were never randomized/assigned to a condition.
Period: Overall Study
Arm/Group | tDCS | Sham tDCS
Started | 27 | 27
Completed | 26 | 25
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: N=62 participants completed baselines and were enrolled in the study. Of these, n=8 were never randomized due to randomization occurring on the day of the first stimulation session.
Groups:
- Not Randomized: Participants were randomized at the beginning of their first tDCS session. Enrolled participants who did not attend their first session (n=8) were never randomized.
- Total: Total of all reporting groups
Arm/Group | tDCS | Sham tDCS | Not Randomized | Total
Number analyzed (Participants) | 27 | 27 | 8 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.19 (7.44) | 34.48 (7.91) | 35.75 (10.38) | 34.08 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 2 | 25
  Male | 18 | 13 | 6 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 0 | 7
  Not Hispanic or Latino | 23 | 24 | 8 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 23 | 22 | 5 | 50
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 8 | 62
Opioid Craving [Mean (Standard Deviation); unit: units on a scale] — Modified Penn Alcohol Craving for Opioids. This measure is self-administered.
  units on a scale | 11.07 (8.39) | 8.85 (7.84) | 8.75 (8.88) | 9.81 (8.12)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Craving
Description: Penn Alcohol Craving (Modified for Opioids). This is a 5-item measure, with each item scored 0 to 6. Items are summed for a total score from 0 to 30. Higher scores = more craving.
Time Frame: 2 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS | Sham tDCS
Number analyzed (Participants) | 26 | 25
units on a scale | 8.92 (1.10) | 8.32 (1.12)
Statistical Analysis 1: Comparison: tDCS vs Sham tDCS; Test type: Superiority; p = .008, Regression, Linear; Utilizing a regression model, baseline craving scores, group condition, and their interaction are regressed on 2-week craving scores; Slope = -.53, 95% CI 2-sided [-.91 to -.15], Standard Error of Mean .190

2. Secondary Outcome: EEG Theta Brainwave Activity
Description: Theta event rate is examined as the number of times/second that brainwaves within the theta frequency range (4-7 Hz). Higher event rates reflect more activity during working memory task.
Time Frame: 2 weeks
Population: theta burst rate (per second) during the 2-back delay part of the working memory task
Measure: Mean (Standard Deviation); unit: events per second
Arm/Group | tDCS | Sham tDCS
Number analyzed (Participants) | 22 | 20
events per second | .38 (.06) | .33 (.05)
Statistical Analysis 1: Comparison: tDCS vs Sham tDCS; Test type: Superiority — An ancova model was conducted comparing differences between tDCS and sham on post-stimulation theta burst rate, while controlling for pre-stimulation theta burst rate; p = .005, ANCOVA

ADVERSE EVENTS:
Time Frame: 2-weeks
Arm/Group | tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 1/27 | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS (N=27) | Sham tDCS (N=27)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Head Itchiness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03842137/Prot_SAP_ICF_000.pdf